CLINICAL TRIAL: NCT07280819
Title: The Impact of Protein Source and Neuromuscular Electrical Stimulation on Muscle Protein Synthesis During Bed Rest
Brief Title: Nutritional and Physical Intervention During Bed Rest
Acronym: Bed-Plant
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Maastricht University Medical Center (Other)
Collaborators: Danone Global Research & Innovation Center (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Basic Science
Other Study IDs: METC 25-020
Record Dates: First submitted 2025-11-20; First posted 2025-12-12 (Actual); Last update posted 2025-12-12 (Actual); Status verified 2025-10

CONDITIONS: Muscle Protein Synthetic Response to Protein
Keywords: muscle biopsy; tracer methodology; NMES

STUDY DESIGN:
Intervention Model Description: The study is a prospective, randomized, parallel-group, controlled interventional trial.
Who Masked: Participant
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Plant-dominant proteins (Experimental)
  Interventions: Dietary Supplement: Nutritionally complete tube feed providing a sole source of nutrition with a plant-dominant protein mix; Device: Neuromuscular Electrical Stimulation (NMES)
- Animal-based proteins (Active Comparator)
  Interventions: Dietary Supplement: Nutritionally complete tube feed providing a sole source of nutrition with an animal-based protein mix; Device: Neuromuscular Electrical Stimulation (NMES)

INTERVENTIONS:
Dietary Supplement: Nutritionally complete tube feed providing a sole source of nutrition with a plant-dominant protein mix — Containing plant-based proteins.
  Arms: Plant-dominant proteins
Dietary Supplement: Nutritionally complete tube feed providing a sole source of nutrition with an animal-based protein mix — Containing animal-based proteins.
  Arms: Animal-based proteins
Device: Neuromuscular Electrical Stimulation (NMES) — The protocol will consist of a warm-up period (5 min), a stimulation period (30min), and a cooling-down period (5min).

SUMMARY:
Hospitalization often involves long periods of bed rest and reduced nutritional intake, which can lead to skeletal muscle loss and anabolic resistance. These effects slow recovery and increase the risk of complications, long-term disability and healthcare costs. Animal-based proteins are effective at stimulating muscle protein synthesis (MPS) because they contain all essential amino acids and have high bioavailability, but they are less sustainable. Plant-based proteins are more environmentally friendly but may be less effective for MPS due to lower essential amino acid content and lower digestibility. Combining different plant proteins may improve their quality, yet their impact during bed rest is still unclear. Neuromuscular electrical stimulation (NMES) may help counteract anabolic resistance by mimicking exercise, but its long-term effects in bedridden individuals are not well studied.

This prospective, randomized, controlled trial aims to assess the effects of a nutritional intervention (plant-dominant versus dairy-based protein) and a physical stimulus (NMES versus non-NMES) on MPS during 4 days of bed rest in healthy young adults.

ELIGIBILITY:
Inclusion Criteria:

* Healthy (assessed based on routine medical questionnaire)
* Male and female sexes
* Aged between 18 and 35 years inclusive
* BMI between 18.5 and 30.0 kg/m²

Exclusion Criteria:

* Vegan diet
* Allergies or intolerance to cow's milk products, fish, soy, and/or pea protein
* Galactosemia
* Smoking on a weekly basis (i.e., every week)
* Diagnosed diabetes mellitus
* Chronic corticosteroid use
* Severe kidney and/or liver failure
* Dialysis
* Bleeding disorders, including anticoagulant and antiplatelet therapy
* Currently pregnant

Ages: 18 Years to 35 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 20 (Estimated)
Dates: Start 2026-01 (Estimated); Primary Completion 2028-01 (Estimated); Study Completion 2029-01 (Estimated)

PRIMARY OUTCOMES:
Muscle protein synthesis rate | 1-4 days
  Muscle protein synthesis rate after 4 day exclusive enteral tube feeding that is nutritionally complete with plant-dominant proteins versus animal-based proteins. This is measured using the deuterated water (2H2O) method.

SECONDARY OUTCOMES:
Muscle protein synthesis rate | 1-4 days
  Muscle protein synthesis rate after NMES versus non-NMES. This is measured using the deuterated water (2H2O) method.
Muscle fiber size in µm² | Final intervention day (after 4 days of enteral feeding and 4 days of NMES)
  Muscle fiber size will be assessed using immunofluorescence staining.
Proportion (%) of muscle fiber types (type I and type II) | Final intervention day (after 4 days of enteral feeding and 4 days of NMES)
  Fiber proportion will be assessed using immunofluorescence staining.
Myonuclei quantity | Final intervention day (after 4 days of enteral feeding and 4 days of NMES)
  Myonuclei quantity will be assessed using immunofluorescence staining.
Mitochondrial Respiratory Capacity in Human Skeletal Muscle Assessed by High-Resolution Respirometry | Final intervention day (after 4 days of enteral feeding and 4 days of NMES)
  Mitochondrial respiratory capacity will be quantified in skeletal muscle fibers using high-resolution respirometry (Oroboros O2k FluoRespirometer). Measurements will include oxygen flux rates across defined respiratory states.

OTHER OUTCOMES:
Age in years | Baseline
  Heteroanamnesia
Body mass in kg | Baseline
  Heteroanamnesia
Height in m | Baseline
  Heteroanamnesia
BMI in kg/m² | Baseline
  Calculated from height and body mass

CONTACTS AND LOCATIONS:
Locations (1):
- Maastricht University, Maastricht, Netherlands

IPD SHARING:
Plan to Share IPD: No